CLINICAL TRIAL: NCT02388633
Title: Acute Microvascular Changes With LDL Apheresis
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Other Study IDs: LDL Apheresis
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Plasmapharesis: Patients undergoing apheresis for elevated LDL. Patients will undergo contrast ultrasound perfusion imaging at rest and during forearm exercise at before and immediately after apheresis.
  Interventions: Procedure: Plasmapharesis

INTERVENTIONS:
Procedure: Plasmapharesis — Clinically-indicated LDL apheresis

SUMMARY:
Severe hypercholesterolemia produced by conditions such as heterozygous familial hypercholesterolemia is associated with multiple complications including premature atherosclerotic disease. There is evidence that microvascular perfusion, particularly flow reserve, in critical organs is limited due to abnormalities in plasma viscosity, abnormal RBC deformability, and an imbalance between vasodilators and vasoconstrictors. There is little is currently known about acute changes in microvascular blood flow and microvascular rheology that occur in response to plasmapharesis which is used in some patients to lower critically elevated cholesterol levels. Our research group has pioneered CEU methods for assessing myocardial and skeletal muscle perfusion, and has previously demonstrated in pre-clinical models that acute hyperlipidemia produces a reduction in microvascular RBC transit rate. In this study, the investigators will assess acute changes in microvascular perfusion in patients undergoing clinically-indicated plasmapharesis.

DETAILED DESCRIPTION:
Subjects who are scheduled to have planned apheresis treatment for severe hypercholesterolemia will be recruited into the study. They will undergo a screening evaluation, including a medical history, physical examination, ECG, and limited echocardiogram to evaluate for exclusion criteria. Before the apheresis procedure, blood samples will be obtained for plasma markers of inflammation, erythrocyte deformability, and plasma viscosity. Contrast enhanced ultrasound perfusion imaging will be performed to evaluate blood flow in the myocardium at rest, as well as in the forearm skeletal muscle before and after mild isometric exercise (50% maximal grip, 0.2 Hz). Flow mediated vasodilation will be performed. The subjects will then undergo their planned apheresis procedure. Within 2 hours of completion of apheresis, blood collection and CEU will be repeated. Plasma lipids will be available as part of the standard apharesis protocol.

ELIGIBILITY:
Inclusion Criteria:

* hypercholesterolemia (LDL >200 mg/dL)
* clinically-indicated aphersis for hyperlipidemia
* age >18 y.o.

Exclusion Criteria:

* pregnant or lactating females
* hypersensitivity to ultrasound contrast agents
* evidence for right to left or bidirectional shunt
* on anticoagulants

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hyperlipidemia undergoing clinically indicated LDL apheresis
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lindner, MD, Principal Investigator — OSHU
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Wu MD, Moccetti F, Brown E, Davidson BP, Atkinson T, Belcik JT, Giraud G, Duell PB, Fazio S, Tavori H, Tsimikas S, Lindner JR. Lipoprotein Apheresis Acutely Reverses Coronary Microvascular Dysfunction in Patients With Severe Hypercholesterolemia. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 1):1430-1440. doi: 10.1016/j.jcmg.2018.05.001. Epub 2018 Jun 19. PMID 29909101

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plasmapharesis
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Plasmapharesis
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Perfusion at Rest
Description: Acoustic intensity data were fit to the following function: y = A(1-e^-beta*t) where y is signal intensity at time t, A is the plateau intensity reflecting relative microvascular blood volume (MBV), and beta is the rate constant reflecting microvascular blood flux rate. Microvascular blood flow was quantified by the product of MBV and beta
Time Frame: 10 min
Measure: Mean (Standard Deviation); unit: IU/s
Arm/Group | Plasmapharesis
Number analyzed (Participants) | 8
IU/s
  Pre-apheresis | 55 (21)
  Post apheresis | 135 (65)

2. Primary Outcome: Skeletal Muscle Perfusion at During Exercise
Description: Contrast ultrasound assessment of microvascular perfusion of forearm skeletal muscle during contractile exercise.
Time Frame: 10 min
Measure: Median (95% Confidence Interval); unit: IU/s
Arm/Group | Plasmapharesis
Number analyzed (Participants) | 8
IU/s
  Pre-apheresis | 116 [76 to 188]
  Post apheresis | 118 [52 to 249]

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Plasmapharesis
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02388633/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02388633/ICF_001.pdf